CLINICAL TRIAL: NCT00103701
Title: Phase I Study of BMS-354825 in Patients With Chronic Accelerated, or Blast Phase Chronic Myelogenous Leukemia or Philadelphia Positive Acute Lymphoblastic Leukemia
Brief Title: BMS-354825 in Patients With Chronic Accelerated, or Blast Phase Chronic Myelogenous Leukemia or Philadelphia Positive Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-002
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Leukemia, Myeloid, Chronic-phase; Leukemia, Lymphoblastic, Acute, Philadelphia-positive
Keywords: Chronic myelogenous leukemia (CML) chronic, accelerated, blast phase; Philadelphia chromosome positive acute (Ph+ALL)
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Bronchiolitis Obliterans Syndrome; Blast Crisis | interventions — Dasatinib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 15- 240 mg, Once or twice daily, 0-3 years depending on response.
  Other Names: Sprycel

SUMMARY:
The purpose of this clinical research study is to understand the safety and efficacy of BMS-354825 in patients with chronic, accelerated, or blast phase chronic myelogenous leukemia (CML) or Philadelphia positive acute lymphoblastic leukemia (ALL) who are resistant to or intolerant of imatinib mesylate (Gleevec).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia chromosome positive, chronic, accelerated or blast phase BML or ALL.
* Patients must have primary or acquired hematologic resistance to imatinib mesylate or have intolerance of imatinib mesylate.
* Men and women, 14 years of age or older.
* Adequate renal function.
* Adequate hepatic function.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month before and at least 3 months after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Patients who are eligible and willing to undergo transplantation during the screening period.
* Women who are pregnant or breastfeeding.
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy.
* Uncontrolled or significant cardiovascular disease.
* Medications that increase bleeding risk.
* Medications that change heart rhythms.
* Dementia or altered mental status that would prohibit the understanding of rendering of informed consent.
* History of significant bleeding disorder or unrelated to CML.
* Evidence of organ dysfunction or digestive dysfunction that would prevent administration of study therapy.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Establishment of MTD and recommended Phase II dose.

SECONDARY OUTCOMES:
1) Hematologic Response 2) Cytogenetic Response.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution, Los Angeles, California
  - Local Institution, Houston, Texas